CLINICAL TRIAL: NCT01124162
Title: Randomized, 2-way Crossover, Bioequivalence Study of Losartan 100 mg Tablets and Cozaar® Administered as 1 * 100 mg Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Losartan 100 mg Tablets in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 30272
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Results first posted 2010-07-19 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic Test Product (Experimental): Losartan 100mg Tablets
  Interventions: Drug: Losartan
- Reference Listed Drug (Active Comparator): Cozaar® 100 mg Tablets
  Interventions: Drug: Cozaar®

INTERVENTIONS:
Drug: Losartan — 100 mg Tablet
  Arms: Generic Test Product
Drug: Cozaar® — 100 mg Tablet
  Other Names: Losartan (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of losartan 100 mg tablets (test) versus Cozaar® (reference), administered as 1 * 100 mg tablet under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Non-child-bearing potential female or male.
* Non-smoker.
* 18 years of age and older.
* Capable of consent.
* Non-child-bearing potential female subject:

  * Post-menopausal state: absence of menses for 12 months prior to drug administration.
  * Surgically sterile: hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to drug administration.

Exclusion Criteria:

* Clinically significant illness within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 100 or over 140 mmHg, diastolic blood pressure lower than 60 or over 100 bpm) at screening.
* Subjects with BMI > 30.0.
* History of significant alcohol abuse within 6 months prior to screening visit or any indication of the regular use of more than 14 units of alcohol per week (1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to the screening visit.
* History of allergic reactions to losartan or other related drugs.
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit drug metabolism within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowl diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the study drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within 90 days preceding study drug administration.
* Any food allergy, intolerance, restriction, or special diet that could, in the opinion of the Medical Sub-Investigator, contraindicate the subjects participation in this study.
* A dept injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood prior to administration of the study medication as follows:

  * Less than 300 mL of whole blood within 30 days
  * 300 mL to 500 mL of whole blood within 45 days, or
  * more than 500 mL of whole blood within 56 days prior to drug administration.
* Consumption of food or beverages containing grapefruit (e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* Clinically significant history of known active hypotension or volume depletion.
* Intolerance to venipuncture.
* Clinically significant history of renal, hepatic, or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis, or glaucoma will not be eligible for this study.
* Subjects unable to understand or unwilling to sign the Informed Consent Form.
* Additional exclusion criteria for females only;

  * Breast-feeding subjects.
  * Positive urine pregnancy test at screening (performed for all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan (Test) First: 100 mg Losartan Tablets test product dosed in first period followed by 100 mg Cozaar® Tablets reference product dosed in the second period.
- Cozaar® (Reference) First: 100 mg Cozaar® Tablets reference product dosed in first period followed by 100 mg Losartan Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Losartan (Test) First | Cozaar® (Reference) First
Started | 40 | 40
Completed | 38 | 40
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Washout of 7 Days
Arm/Group | Losartan (Test) First | Cozaar® (Reference) First
Started | 38 | 40
Completed | 37 | 40
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Losartan (Test) First | Cozaar® (Reference) First
Started | 37 | 40
Completed | 37 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan (Test) First | Cozaar® (Reference) First | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 31 | 31 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black | 1 | 1 | 2
  Caucasian | 32 | 36 | 68
  Hispanic | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Losartan (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Losartan Cmax.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Losartan: 100 mg Losartan Tablets test product dosed in either period.
- Cozaar®: 100 mg Cozaar® Tablets reference product dosed in either period.
Arm/Group | Losartan | Cozaar®
Number analyzed (Participants) | 77 | 77
ng/mL | 637.01 (340.35) | 582.39 (327.20)
Statistical Analysis 1: Comparison: Losartan vs Cozaar®; Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level; Ratio of the T/R geometric mean x 100 = 108.14, 90% CI 2-sided [97.43 to 120.03] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Losartan (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Losartan AUC0-t.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan | Cozaar®
Number analyzed (Participants) | 77 | 77
ng*h/mL | 950.90 (422.61) | 934.24 (418.99)
Statistical Analysis 1: Comparison: Losartan vs Cozaar®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101.70, 90% CI 2-sided [98.57 to 104.93] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Losartan (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Losartan AUC0-inf.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan | Cozaar®
Number analyzed (Participants) | 77 | 77
ng*h/mL | 962.67 (423.97) | 947.18 (419.38)
Statistical Analysis 1: Comparison: Losartan vs Cozaar®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101.5, 90% CI 2-sided [98.41 to 104.68] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax of Losartan Carboxy Acid (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Informational comparison of Cmax values for the metabolite Losartan Carboxy Acid.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Losartan | Cozaar®
Number analyzed (Participants) | 77 | 77
ng/mL | 658.17 (272.35) | 647.22 (259.27)
Statistical Analysis 1: Comparison: Losartan vs Cozaar®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.08, 90% CI 2-sided [98.24 to 106.06] — This analysis was for informational purposes only and was not used to establish bioequivalence

5. Secondary Outcome: AUC0-t of Losartan Carboxy Acid (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Informational comparison of AUC0-t values for the metabolite Losartan Carboxy Acid.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan | Cozaar®
Number analyzed (Participants) | 77 | 77
ng*h/mL | 3748.87 (1314.68) | 3750.39 (1312.04)
Statistical Analysis 1: Comparison: Losartan vs Cozaar®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.31, 90% CI 2-sided [97.84 to 102.84] — This analysis was for informational purposes only and was not used to establish bioequivalence

6. Secondary Outcome: AUC0-inf of Losartan Carboxy Acid(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Informational comparison of AUC0-inf values for the metabolite Losaran Carboxy Acid.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan | Cozaar®
Number analyzed (Participants) | 77 | 77
ng*h/mL | 3855.02 (1345.50) | 3858.92 (1352.83)
Statistical Analysis 1: Comparison: Losartan vs Cozaar®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.25, 90% CI 2-sided [97.87 to 102.69] — This analysis was for informational purposes only and was not used to establish bioequivalence

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 2 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Losartan | Cozaar®
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 14/80 | 9/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=80) | Cozaar® (N=80)
Low Blood Pressure (General disorders) | 7 (7) | 3 (5)
Headache (General disorders) | 5 (6) | 3 (4)
Dizziness (General disorders) | 3 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.